CLINICAL TRIAL: NCT05646615
Title: Experiences and Health-related Quality of Life of Informal Caregivers of Patients Who Start Home Dialysis: a Prospective, Multicenter Cohort Study
Brief Title: Experiences and Health-related Quality of Life of Informal Caregivers of Dialysis Patients
Status: Completed | Type: Observational
Sponsor: B.C. van Jaarsveld (Other)
Collaborators: Admiraal de Ruyter Hospital (Other); Alrijne Hospital (Other); Amphia Hospital (Other); St. Antonius Hospital (Other); Canisius-Wilhelmina Hospital (Other); Catharina Ziekenhuis Eindhoven (Other); Deventer Ziekenhuis (Other); Dialysis Center Beverwijk (Unknown); Tergooi Hospital (Other); Diapriva Dialysis Center, Amsterdam (Other); Elkerliek Hospital (Other); Flevoziekenhuis (Other); Gelre Hospitals (Other); Groene Hart Ziekenhuis (Other); Haga Hospital (Other); Isala (Other); Laurentius Hospital (Unknown); Maasstad Hospital (Other); Maxima Medical Center (Other); Noordwest Ziekenhuisgroep (Other); OLVG Oost (Unknown); OLVG West (Unknown); Radboud University Medical Center (Other); Reinier de Graaf Groep (Other); Rijnstate Hospital (Other); Saxenburgh Group (Unknown); Slingeland Hospital (Other); UMC Utrecht (Other); VieCuri Medical Centre (Other); Amsterdam UMC (Other); Bernhoven Hospital (Other); ZorgSaam (Unknown); Jessa Hospital (Other)
Responsible Party: Sponsor-Investigator, B.C. van Jaarsveld, Principal Investigator, Amsterdam UMC, location VUmc
Organization: Amsterdam UMC, location VUmc (Other)
Other Study IDs: 21OM+003
Record Dates: First submitted 2022-11-21; First posted 2022-12-12 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Peritoneal Dialysis; Hemodialysis, Home; Hemodialysis; Quality of Life; Informal Caregivers; Family Caregivers; Renal Replacement Therapy; Kidney Failure, Chronic; Patient Reported Outcome Measures
Keywords: End-Stage Kidney Disease; Informal Caregivers; Quality of Life; Experiences
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this prospective, observational, multicentre cohort study is to assess the trajectory of the experiences (both positive and negative) and health-related quality of life (HRQOL) of informal caregivers of patients who start home dialysis, and compare these to experiences and HRQOL of informal caregivers of patients who start in-centre hemodialysis. The investigators hypothesise that informal caregivers of home dialysis patients experience more positive experiences, but also more negative experiences, and still have better HRQoL, compared with caregivers of in-centre HD patients. Participants will fill in five different validated questionnaires and questions on required support. Participants are asked to fill in the questionnaires after inclusion (i.e., start of dialysis), and at 6 and 12 months after start dialysis.

DETAILED DESCRIPTION:
End-stage kidney disease, the need to start dialysis, and the choice for a home-based treatment or a centre-based treatment does not only have an effect on patients, but also on their informal caregivers like spouses and adult children providing care to the patient. In order to properly inform patients with end-stage kidney disease and their informal caregivers about the start of dialysis therapy and the choice of dialysis modality, it is important to discuss also what the caregiver can expect after the start of dialysis. However, available evidence regarding the course of caregiving experiences after start of dialysis is limited. The aim of this study is to assess the trajectory of the experiences (both positive and negative) and health-related quality of life (HRQoL) of caregivers of patients who start home dialysis, and compare these to experiences and HRQoL of caregivers of patients who start in-centre hemodialysis (HD). The investigators hypothesise that (co-residential) caregivers of home dialysis patients experience more positive experiences, but also more negative experiences, and still have better HRQoL, compared with caregivers of in-centre HD patients.

This study is a prospective, observational, multicentre cohort study which is an extension of the ongoing DOMESTICO study. DOMESTICO is a nationwide study in incident dialysis patients, investigating the effects of home dialysis on HRQoL in relation to clinical outcome and costs, in comparison to in-centre HD. Participants will fill in five different validated questionnaires and questions on required support. Participants are asked to fill in the questionnaires after inclusion (i.e., start of dialysis), and at 6 and 12 months after start dialysis.

ELIGIBILITY:
Inclusion Criteria:

* Informal caregivers who care for a partner, family member, friend or loved one with end-stage kidney disease who is starting dialysis therapy and is included in the DOMESTICO study
* 18 years or older

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Informal caregivers of patients who are starting dialysis and are included in the DOMESTICO study
Sampling Method: Non-Probability Sample
Enrollment: 202 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Changes in positive experiences of the caregiver (PES) | Baseline (start of dialysis), and 6 months and 12 months after start dialysis
  Positive Experiences Scale (PES): a Dutch 8-item validates questionnaire

SECONDARY OUTCOMES:
Changes in negative experiences of the caregiver (EDIZ+) | Baseline (start of dialysis), and 6 months and 12 months after start dialysis
  'Ervaren Druk door Informele Zorg' or Experienced Burden by Informal Care (EDIZ+): a Dutch 15-item validated questionnaire
Changes in negative experiences of the caregiver (CES-D) | Baseline (start of dialysis), and 6 months and 12 months after start dialysis
  Centre for Epidemiologic Studies Depression Scale (CES-D): a 20-item validated questionnaire
Changes in health-related quality of life (HRQOL) (SF-12) | Baseline (start of dialysis), and 6 months and 12 months after start dialysis
  12-item Short Form (SF-12): validated questionnaire with eight domains
Changes in health-related quality of life (HRQOL) (EQ5D-5L) | Baseline (start of dialysis), and 6 months and 12 months after start dialysis
  EuroQol-5D-5L (EQ5D-5L): validated questionnaire with five domains

OTHER OUTCOMES:
Required support | Baseline (start of dialysis), and 6 months and 12 months after start dialysis
  Exploratory outcome, assessed by a questionnaire investigating in which domains caregivers would like extra support

CONTACTS AND LOCATIONS:
Overall Officials: Brigit C van Jaarsveld, MD, PhD, Principal Investigator — Amsterdam UMC, location VUmc
Locations (33):
- Jessa Hospital, Hasselt, Belgium
- Netherlands (32):
  - Noordwest Ziekenhuisgroep, Alkmaar
  - Flevoziekenhuis, Almere Stad
  - Alrijne Hospital, Alphen aan den Rijn
  - Amsterdam UMC, Amsterdam
  - Diapriva Dialysis Center, Amsterdam
  - OLVG Oost, Amsterdam
  - OVLG West, Amsterdam
  - Gelre Hosptials, Apeldoorn
  - Rijnstate Hospital, Arnhem
  - Dialysis Center Beverwijk, Beverwijk
  - Amphia Hospital, Breda
  - Reinier de Graaf Group, Delft
  - Deventer Hospital, Deventer
  - Slingeland Hospital, Doetinchem
  - Catharina Hospital, Eindhoven
  - Admiraal de Ruyter Hospital, Goes
  - Groene Hart Hospital, Gouda
  - Saxenburgh Group, Hardenberg
  - Elkerliek Hospital, Helmond
  - Dialysis Center Tergooi, Hilversum
  - Antonius Hospital, Nieuwegein
  - Canisius-Wilhelmina Hospital, Nijmegen
  - Radboudumc, Nijmegen
  - Laurentius Hospital, Roermond
  - Maasstad Hospital, Rotterdam
  - ZorgSaam, Terneuzen
  - Haga Hospital, The Hague
  - Bernhoven Hospital, Uden
  - UMC Utrecht, Utrecht
  - Maxima Medical Center, Veldhoven
  - VieCuri Medical Center, Venlo
  - Isala Hospital, Zwolle

IPD SHARING:
Plan to Share IPD: No